CLINICAL TRIAL: NCT02348515
Title: Effects of ACE2/Ang-(1-7) on Cardiac Progenitor Cells From Heart Failure Patients and Explant Control
Brief Title: Cardiovascular Disease Protection Tissue
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201300122-N; R01HL056921 (NIH)
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and discarded heart tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Heart failure or coronary disease: This group will have small samples collected from the apex core (that would be routinely discarded at the time of the implantation procedure) by undergoing a left ventricular assist device implantation. In addition, a blood sample will be collected.
  Interventions: Procedure: Heart failure or coronary disease; Procedure: Blood Draw
- Heart transplant patients: This group will have multiple samples collected including, excess myocardial biopsy samples that will not be utilized by pathology. In addition, a blood sample will be collected.
  Interventions: Procedure: Heart transplant patients; Procedure: Blood Draw
- Orthotopic Heart Transplant Patients: This group will have myocardial tissue samples collected from the diseased heart. In addition, a blood sample will be taken.
  Interventions: Procedure: Orthotopic Heart Transplant Patients; Procedure: Blood Draw
- Heart Surgery Patients: This groups will have samples collected from the left atrial appendages that are routinely removed to prevent thrombosis during atrial fibrillation surgery and a piece of the right atria will be cut in order to implant the cannula. In addition, a blood sample will be taken.
  Interventions: Procedure: Heart Surgery Patients; Procedure: Blood Draw

INTERVENTIONS:
Procedure: Heart failure or coronary disease — Small samples collected from the apex core in the heart. In addition, blood samples will be taken.
  Groups: Heart failure or coronary disease
Procedure: Heart transplant patients — Heart samples collected including, excess myocardial biopsy samples. In addition, blood samples will be taken.
  Groups: Heart transplant patients
Procedure: Orthotopic Heart Transplant Patients — Myocardial tissue samples collected from the diseased heart. In addition, blood samples will be taken.
  Groups: Orthotopic Heart Transplant Patients
Procedure: Heart Surgery Patients — Heart samples will be collected from the left atrial appendages. In addition, blood samples will be taken.
  Groups: Heart Surgery Patients
Procedure: Blood Draw — All subjects will have 20 ml of blood drawn for further analysis.

SUMMARY:
Recent evidence of a potential role for cardiac progenitor cells (CPCs) in cardiac repair and the discovery of a vasoprotective axis of the renin-angiotensin system (RAS) offer such breakthroughs. Investigators have observed that an imbalance in the vasoprotective axis {angiotensin converting enzyme 2 (ACE2)/angiotensin-(1-7) [Ang-(1-7)]/Mas receptor} and the vasodeleterious axis [angiotensin converting enzyme (ACE)/angiotensin II (AngII)/AngII type 1 receptor (AT1R)] of the RAS within the CPCs affects their functionality and regenerative potential. Investigators believe that restoring the balance between these two axes of the RAS is essential to improve CPC function and enhance their reparative capabilities. These observations have led to the hypothesis that genetic modification of CPCs by overexpression of ACE2/Ang-(1-7) will enhance their reparative function and improve their potential to attenuate myocardial ischemia-induced cardiac damage.

DETAILED DESCRIPTION:
As a participant undergoes a clinically indicated heart transplant, or a left ventricular assist device (LVAD) implantation, or a right heart biopsy, or atrial fibrillation surgery, or right atria cannulation, the following tissue samples will be collected:

In the subjects undergoing orthotopic heart transplant (n=20), failed myocardial tissue samples will be collected from the diseased heart.

For subjects undergoing left ventricular assist device implantation (n=60), small samples will be collected from the apex core (that would be routinely discarded at the time of the implantation procedure).

For heart transplant subjects undergoing clinically indicated right heart biopsy (n=20), the collection of multiple samples including, excess myocardial biopsy samples that will not be utilized by pathology.

For subjects undergoing any heart surgery (n=80), the collection of left atrial appendages that are routinely removed to prevent thrombosis during atrial fibrillation surgery and a piece of the right atria will be cut in order to implant the cannula.

In addition, a collection of 20ml (about one tablespoon) of blood will be taken from all subjects to analyze progenitor/inflammatory cells and inflammation cytokines and pertinent medical history.

ELIGIBILITY:
Inclusion Criteria:

* heart transplant surgery
* left ventricular assist device implantation
* heart surgery required for atrial fibrillation and right atria cannulation

Exclusion Criteria:

* We are collecting discarded tissues following surgery. There is no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing orthotopic heart transplant, left ventricular assist device implantation, right heart biopsy, and any other heart surgery (atrial fibrillation and right atria cannulation).
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-06; Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Imbalance of vasoprotective and vasodeleterious axes of the renin angiotensin system (RAS) is associated with dysfunction of CPC isolated from diseased tissue | two years
  CPCs will be isolated from the collected heart tissue. Function assay such as proliferation, migration, reactive oxygen species (ROS) level will be analyzed. Renin-angiotensin system (RAS) genes and inflammatory cytokines will be quantifies using polymerase chain reaction (PCR) and protein assay to investigate if the cell dysfunction is associated with the imbalance of vasoprotective and vasodeleterious axes of the RAS.

SECONDARY OUTCOMES:
Screening for biomarkers related to clinic outcome in the blood | two years
  Progenitor/inflammatory cells, inflammatory cytokines, and growth factors will be measured to determine if they are associated with heart diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Pepine, MD, Principal Investigator — University of Florida
Locations (1):
- Yanfei Qi, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No